CLINICAL TRIAL: NCT03553303
Title: Pharmacodynamic Effects of Sacubitril/Valsartan on Natriuretic Peptides, Angiotensin and Neprilysin. A Ringerike Heart Failure Cohort Phase IV Study of Angiotensin Receptor Neprilysin Inhibiton
Brief Title: Pharmacodynamic Effects of Sacubitril/Valsartan on Natriuretic Peptides, Angiotensin and Neprilysin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Christian Hall, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3403003
Record Dates: First submitted 2018-05-23; First posted 2018-06-12 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Increasing doses of Sacubitril/Valsartan
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet — Increasing doses of Sacubitril/Valsartan

SUMMARY:
The study measure multiple neurohormones in patients with heart failure being treated with Sacubitril/Valsartan in increasing doses over an 8 week period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written informed consent before any study assessment is performed.
2. Ambulatory ≥ 18 years of age, male or female, treated at Ringerike Hospital.
3. Patients with symptomatic chronic heart failure and reduced ejection fraction (≤ 40%).
4. Patients on optimized medical treatment for heart failure. -

Exclusion Criteria:

1. Patients not able to comply in the study.
2. Patients having contraindication for treatment with Entresto;

   1. Hypersensitivity to the active substances or to any of the excipients listed in section
   2. Hyperkalemia: > 5.4 mmol/L
   3. Known history of angioedema related to previous ACE inhibitor or ARB therapy.
   4. Hereditary or idiopathic angioedema.
   5. Concomitant use with Aliskiren-containing medicinal products in patients with diabetes mellitus or in patients with renal impairment (eGFR <60 ml/min/1.73m2)
   6. End-stage renal disease (<15 mL/min per 1.73m2 or treatment by dialysis).
   7. Severe hepatic impairment, biliary cirrhosis and cholestasis (Child-Pugh C classification).
   8. Pregnancy Breast-feeding-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Neurohormonal plasma concentration | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hall, MD PhD, Study Chair — University of Oslo
Locations (1):
- Ringerike Hospital Vestre Viken Hospital Trust, Hønefoss, Buskerud, Norway

IPD SHARING:
Plan to Share IPD: No